CLINICAL TRIAL: NCT04863131
Title: Safety and Immunogenicity of Intradermal SARS-CoV-2 Vaccine EXG-5003 in Healthy Adults
Brief Title: Safety and Immunogenicity of EXG-5003
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fujita Health University (Other)
Collaborators: Elixirgen Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Yohei Doi, Professor and Chair of the Department of Microbiology, Fujita Health University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EXG-5003-J01
Record Dates: First submitted 2021-04-15; First posted 2021-04-28 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXG-5003 (Experimental)
  Interventions: Biological: EXG-5003
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: EXG-5003 — COVID-19 self-replicating mRNA vaccine
  Arms: EXG-5003
Biological: Placebo — placebo solution
  Arms: Placebo

SUMMARY:
This is a First in Human, randomized, placebo-controlled Phase I/II trial to evaluate the safety and immunogenicity of the intradermal COVID-19 vaccine, EXG-5003 in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Has provided written consent for participation
* Age between 20 and 55
* Has a negative nucleic acid-based test result for SARS-CoV-2
* Has a negative antibody test result for SARS-CoV-2

Exclusion Criteria:

* Signs and symptoms consistent with COVID-19 upon screening
* History of COVID-19
* Presence of uncontrolled cardiovascular, hematologic, respiratory, hepatic, renal, gastrointestinal, or neuropsychiatric disease
* Presence of diabetes mellitus
* Presence of active autoimmune disease
* Positive for HBc, HCV or HIV antibody
* History of anaphylactic shock
* History of epilepsy
* Presence of active malignancy
* Presence of lung disease (e.g., COPD, asthma)
* Positive urine pregnancy test within 24 hours
* Pregnant, lactating, planned pregnancy of self (if female) or partner (if male) within 90 days after administration of the trial drug
* If female and premenopausal, not agreeable to contraception for 90 days after second administration of the trial drug
* If male, not agreeable to contraception for 90 days after second administration of the trial drug
* Presence of clinically relevant electrocardiogram or vital sign abnormality at screening
* Participated in a clinical trial of a drug or a medical device within 30 days or a biologic within 90 days
* Received any SARS-CoV-2 vaccine
* Received within 90 days, or is planning to receive during the study period, an immunoglobulin or blood product
* Received within 180 days, or is planning to receive during the study period, a biologic product with immunosuppressive properties
* Received for 14 days or more within 180 days, or is planning to receive during the study period, a corticosteroid
* Deemed ineligible for the study as determined by the principal investigator or a co-investigator

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants Reporting Local and Systemic Adverse Events | Day 1 up to Day 365 post dose

SECONDARY OUTCOMES:
Flowcytometry assay to enumerate the frequency of T cells expressing CD3, CD4, CD8, CD62L, CD45RA, IFN-γ, IL-4, CD107, TNF, IL-2, IL-6, CD154 (CD40L), Perforin, and Granzyme B. | Day15, Day29, Day43, Day57, Day92, Day183, Day365
Assessment of T cells by Intracellular cytokine staining assays | Day15, Day29, Day57,
Genometric Mean Titer (GMT) of serum anti-RBD IgG | Day15, Day29, Day43, Day57, Day92, Day183, Day365
GMT of neutralizing antibody | Day15, Day29, Day43, Day57, Day92, Day183, Day365

CONTACTS AND LOCATIONS:
Overall Officials: Yohei Doi, MD, Principal Investigator — Fujita Health University Hospital
Locations (1):
- Fujita Health University Hospital, Toyoake, Aichi-ken, Japan